CLINICAL TRIAL: NCT03926767
Title: Additional Effect of Pain Neuroscience Education to Orofacial Manual Therapy and Orofacial and Neck Motor Control Exercises for Pain Intensity and Disability in Temporomandibular Disorders: a Randomized Clinical Trial
Brief Title: Additional Effect of Pain Neuroscience Education to Orofacial and Neck Exercises in Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3449/2018
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Disorders
Keywords: Pain Neuroscience Education; Chronic Pain; Orofacial Manual Therapy; Orofacial exercises; Neck Motor Control Exercises
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education + orofacial and neck exercises (Experimental): All participants in this arm will initially receive two additional sessions in which a workshop on PNE will be administered and discussed. A power-point presentation with metaphors and animated videos will be employed. The PNE program will be held in 2 sessions of 30 minutes each. A protocol of Orofacial Exercises and Manual Therapy will be adopted in the present study. A protocol of neck motor control protocol will be adopted in our study. The exercises will be administered during six weeks, twice a week. One session will run in the outpatient clinic and the other will be home based. Half of the sessions will be comprised of orofacial strategies and the other half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
  Interventions: Other: Pain Neuroscience Education (PNE); Other: Orofacial Manual Therapy; Other: Orofacial Exercises; Other: Neck Motor Control Exercises
- Orofacial and neck exercises (Active Comparator): A protocol of neck motor control protocol will be adopted in our study. The exercises will be administered during six weeks, twice a week. One session will run in the outpatient clinic and the other will be home based. Half of the sessions will be comprised of orofacial strategies and the other half neck motor control exercises. Each exercise and technique will be administered 10 times for 10 seconds.
  Interventions: Other: Orofacial Manual Therapy; Other: Orofacial Exercises; Other: Neck Motor Control Exercises

INTERVENTIONS:
Other: Pain Neuroscience Education (PNE) — A power-point presentation with metaphors and animated videos will be employed. The PNE program will be held in 2 sessions of 30 minutes each. The intervention program will be divided into 17 thematic topics according to Explain Pain.
  Arms: Pain Neuroscience Education + orofacial and neck exercises
Other: Orofacial Manual Therapy — A protocol of Orofacial Exercises and Manual Therapy will be adopted in the present study. The manual therapy techniques will be: Intraoral temporalis release, Intraoral medial and lateral pterygoid (origin) technique and Intraoral sphenopalatine ganglion technique.
Other: Orofacial Exercises — Two mandibular exercises: Mandibular body-condylar cross-pressure chewing technique and Post-isometric relaxation stretches-laterotrusion and opening. Each exercise will be executed 10 times per session for 10 seconds.
Other: Neck Motor Control Exercises — A protocol of neck motor control protocol will be adopted in our study. The exercises included bracing exercises (six hierarchical levels) in neurodevelopment stages for the cervical spine. Extremity range of motion exercises will be conducted while maintaining a stable spine at the specific positions. Also, cervical isometric exercises (five hierarchical levels) will be carried out directly forward, obliquely, toward right and left, and directly backward by maintaining a stable spine with elastic resistive bands. Finally, exercises also included functional training with elastic resistance and exercise balls on unstable surfaces (eight hierarchical levels). The criteria to progress in each exercise domain (bracing, isometric exercises or functional training) will be sustain the contraction for 10 seconds, 10 times.

SUMMARY:
The objective of this study will be to verify the additional effect of Pain Neuroscience Education program to orofacial manual therapy and orofacial and neck motor control exercises for pain intensity and disability and for the secondary outcomes pain self-efficacy, kinesiophobia, and overall perception of improvement in patients with Temporomandibular Disorders (TMD). This study will be a randomized clinical trial comprising a sample of 148 participants. Subjects will undergo a screening process to verify those presenting a diagnosis of painful TMD confirmed by the Research Diagnostic Criteria (RDC/TMD), between 18 and 55 years of both genders, and then the volunteers will be randomized into two groups (G1: Pain Neuroscience Education + Orofacial Manual Therapy/orofacial exercises/neck motor control exercises vs. G2: Orofacial Manual Therapy/orofacial exercises/neck motor control exercises). These volunteers will be recruited at the Dentistry Clinic of the University of São Paulo's School of Dentistry of Ribeirão Preto - University of São Paulo. The intervention will be administered twice a week for 6 weeks by a single therapist lasting 1 hour per session. The primary outcome will be pain intensity and disability and the secondary outcomes will be pain self-efficacy, kinesiophobia and overall perception of improvement. The participants will be assessed immediate after the last session and at one and three-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of painful TMD Research Diagnostic Criteria for TMD (RDC/TMD)
* A history of orofacial pain at least three months prior to the study (TREEDE et al, 2015)
* age ranging between 18 to 55 years, considering the greater prevalence of TMD associated with this age period.

Exclusion Criteria:

* Patients with illiteracy, severe depression (medical diagnoses), clinical history of tumors in the craniofacial region, patients in the post dental surgery period or submitted to previous physical therapy in the past year or to any health/pain education strategy, pregnant women, infections, whiplash-associated disorders and with chronic degenerative inflammatory or neurologic disorders were excluded from this study. Patients will be instructed to not use pain relief medications during the intervention period of this trial and if any medication be used, participants will be encouraged to report.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | Immediately after, one- and three-month follow-up
  The Numerical Pain Rating Scale will be used to assess pain intensity in this trial and consists in a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable".
Change in Orofacial Pain related Disability | Immediately after, one- and three-month follow-up
  The Craniofacial Pain and Disability Inventory (CF-PDI) is a self-administered questionnaire that measures the outcomes of pain and disability related to craniofacial pain and demonstrated a good structure, internal consistency, reproducibility, and construct validity. Also, the Brazilian Portuguese version showed acceptable psychometric measurements. It consists of 21 items, with a score ranging from 0 to 63 points. Each question is scored on 4-point ordinal scale, ranging from 0 to 3. A higher score reflects higher disability levels.

SECONDARY OUTCOMES:
Change in Pain Self-Efficacy Questionnaire (PSEQ) | Immediately after, one- and three-month follow-up
  Study participants will be evaluated on self-efficacy related to chronic pain, which can be defined as an individual's confidence he/she can successfully produce desirable results related to living with chronic pain. The PSEQ has 10 items which are rated on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident"). It was adapted and validated to Brazilian Portuguese (Sarda et al, 2007). Previous research showed an effect on self-efficacy using a PNE intervention based on metaphors compared to an intervention using cognitive-behavioral concepts.
Change in Kinesiophobia | Immediately after, one- and three-month follow-up
  The Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK/TMD) is self-report questionnaire that assesses the fear of movement. In this study, the TSK-TMD with 12 items validated in Brazilian Portuguese was used and showed acceptable psychometric measurements. Each item is scored on a 4-point ordinal scale, ranging from 'strongly disagree' (score = 1) to 'strongly agree' (score = 4). Ratings are summed to yield a total score. Higher scores reflect a greater fear of movement (12-48 points).
Change in Global Perceived Improvement | Immediately after, one- and three-month follow-up
  The global perceived effect (GPE) used for this trial is an 11-point scale that ranges from -5 ("vastly worse") through 0 ("no change") to +5 ("completely recovered") and participants are asked: "Compared to when this episode first started, how would you describe your back these days?". A higher score indicates higher perception of recovery from the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Thais Chaves, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aguiar ADS, Moseley GL, Bataglion C, Azevedo B, Chaves TC. Education-Enhanced Conventional Care versus Conventional Care Alone for Temporomandibular Disorders: A Randomized Controlled Trial. J Pain. 2023 Feb;24(2):251-263. doi: 10.1016/j.jpain.2022.09.012. Epub 2022 Oct 8. PMID 36220481
- [Derived] Dos Santos Aguiar A, Bataglion C, Felicio LR, Azevedo B, Chaves TC. Additional effect of pain neuroscience education to craniocervical manual therapy and exercises for pain intensity and disability in temporomandibular disorders: a study protocol for a randomized controlled trial. Trials. 2021 Sep 6;22(1):596. doi: 10.1186/s13063-021-05532-x. PMID 34488856